CLINICAL TRIAL: NCT07005505
Title: Automatic Tube Compensation vs. Pressure Support Ventilation During Spontaneous Breathing Trials in Critically Ill Adults: A Cluster-Randomized, Cluster-Crossover Trial
Brief Title: Automatic Tube Compensation vs. Pressure Support Ventilation During Spontaneous Breathing Trials in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Jie Li, Professor, Rush University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 25031208
Record Dates: First submitted 2025-05-19; First posted 2025-06-05 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Spontaneous Breathing Trial in ICU
Keywords: Ventilator liberation; Spontaneous breathing trial

STUDY DESIGN:
Intervention Model Description: During the first month of the study, each intensive care unit (ICU) will be randomly assigned to one mode of spontaneous breathing trial (SBT). Each month thereafter, each ICU will independently alternate between the two modes. Patients will be analyzed based on the group to which they were assigned at enrollment (intention-to-treat), even if they remain in the study ICU during a transition from one month to the next or transfer to another ICU assigned to the opposite SBT mode ("crossover"). The last three days of each month will serve as an analytic washout period, during which the study ICU will continue using the assigned ventilator mode, but new patients will not be included in the primary analysis. This three-day washout period is intended to minimize the number of patients experiencing a "crossover" between assigned modes within the 72-hour timeframe used to assess feasibility outcomes and adherence.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adult Intensive Care Unit (AICU) (Experimental)
  Interventions: Other: Pressure Support Ventilation (PSV); Other: Automatic tube compensation (ATC)
- Medical Intensive Care Unit (MICU) (Experimental)
  Interventions: Other: Pressure Support Ventilation (PSV); Other: Automatic tube compensation (ATC)
- Cardiosciences Intensive Care Unit (CSICU) (Experimental)
  Interventions: Other: Pressure Support Ventilation (PSV); Other: Automatic tube compensation (ATC)
- Neuroscience Intensive Care Unit (NSICU) (Experimental)
  Interventions: Other: Pressure Support Ventilation (PSV); Other: Automatic tube compensation (ATC)

INTERVENTIONS:
Other: Pressure Support Ventilation (PSV) — Spontaneous breathing trials will be conducted using the mode pressure support ventilation (PSV) with settings of a pressure support of 5 cmH2O and positive end expiratory pressure (PEEP) 5 cmH2O.
Other: Automatic tube compensation (ATC) — Spontaneous breathing trials will be conducted using the mode automatic tube compensation (ATC) with settings of 100% tube compensation and a positive end expiratory pressure (PEEP) of 5 cmH2O.

SUMMARY:
For patients requiring mechanical ventilation, spontaneous breathing trials (SBTs) are conducted to determine if it is safe to remove the breathing tube. There are multiple methods for conducting SBTs. The purpose of this study is to compare the effects of 2 methods, pressure support ventilation (PSV) versus automatic tube compensation (ATC), on successful extubation for critically ill adult patients who received mechanical ventilation for over 24 hours.

DETAILED DESCRIPTION:
The delivery of pressure support through the ventilator can be fixed using the pressure support ventilation (PSV) mode or variable using the automatic tube compensation (ATC) mode. Similar to PSV, ATC provides pressure support but dynamically adjusts it to compensate the resistive work of breathing and the mechanical load on respiratory muscles imposed by an artificial airway, such as an endotracheal or tracheostomy tube. Although both ATC and PSV are licensed and used in clinical practice, the optimal method to deliver pressure support during a spontaneous breathing trial (SBT) remains unknown. At Rush University Medical Center, ATC has been used for SBTs for over a decade. However, given the growing popularity of PSV, the SBT protocol was updated and now approves the use of PSV and ATC as standard care for SBT without making a recommendation for a preferred mode. The choice between PSV and ATC during SBT is left to the discretion of the clinician, reflecting the ongoing equipoise in the conduct of the SBT. As patients will be exposed to the potential benefits and risks of PSV or ATC under this change in clinical practice, the investigators are conducting a cluster-randomized cluster-crossover trial to compare the mode's effect on successful extubation.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to intensive care unit (ICU)
* Age 18 years or older
* Requiring invasive mechanical ventilation for at least 24 hours
* Pass spontaneous breathing trial screen criteria

Exclusion Criteria:

* Clinical decision made not to proceed with extubation regardless of spontaneous breathing trial (SBT) results
* Do not intubate (DNI) order
* Presence of tracheostomy
* Pregnancy
* Known prisoner
* Immediate need for extubation, self-extubation, or unplanned extubation that precludes safe performance of study procedures
* Enrolled in another clinical trial that impacts ventilator weaning or liberation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Reintubation | Within 48 hours of extubation
Death | Within 48 hours of extubation

SECONDARY OUTCOMES:
Time to successful extubation | From the start of the first spontaneous breathing trial (SBT) to the first successful extubation (without reintubation within 48 hours) or death from any cause, whichever occurred first, assessed up to 30 days.
  The duration (in hours) from the spontaneous breathing trial (SBT) initiation to extubation without reintubation within 48 hours
Spontaneous breathing trial (SBT) results | Up to 30 days from study enrollment or until hospital discharge, whichever occurs first.
  SBT results (pass or fail) for the first 3 attempts if conducted
Reintubation | within 24 hours of extubation
Reintubation | Within 72 hours of extubation
Reintubation | Within 7 days of extubation
Use of noninvasive respiratory support | Within 48 hours of extubation
  Use of noninvasive ventilation, continuous positive airway pressure (CPAP), and high flow nasal cannula (HFNC) and its duration
Total duration of mechanical ventilation | From the date of intubation to the date of extubation without reintubation within 28 hours or date of death from any cause, whichever occurs first, assessed up to 30 days.
Intensive care unit (ICU) length of stay (LOS) | From the date of ICU admission to the date of ICU discharge, assessed up to 30 days.
Hospital length of stay (LOS) | From the date of hospital admission to the date of hospital discharge, assessed up to 30 days.
Mortality | At intensive care unit (ICU) discharge
Mortality | Up to 30 days
Clinician adherence to initially assigned spontaneous breathing trial (SBT) mode | Up to 30 days
Ventilator associated complications | From the date of intubation to the date of extubation without reintubation in 48 hours or death from any cause, whichever occurs first, assessed up to 30 days.
  Including ventilator associated pneumonia, skin pressure ulcers, and barotrauma such as pneumothorax, pneumomediastinum, or subcutaneous emphysema

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Latronico N, Rasulo FA, Eikermann M, Piva S. Illness Weakness, Polyneuropathy and Myopathy: Diagnosis, treatment, and long-term outcomes. Crit Care. 2023 Nov 13;27(1):439. doi: 10.1186/s13054-023-04676-3. PMID 37957759
- [Background] Hoshino T, Yoshida T. Spontaneous breathing-induced lung injury in mechanically ventilated patients. Curr Opin Crit Care. 2025 Feb 1;31(1):5-11. doi: 10.1097/MCC.0000000000001231. Epub 2024 Nov 8. PMID 39526662
- [Background] Li W, Cai J, Ding L, Chen Y, Wang X, Xu H. Incidence and risk factors of ventilator-associated pneumonia in the intensive care unit: a systematic review and meta-analysis. J Thorac Dis. 2024 Sep 30;16(9):5518-5528. doi: 10.21037/jtd-24-150. Epub 2024 Sep 14. PMID 39444919
- [Background] Guerin C, Terzi N, Mezidi M, Baboi L, Chebib N, Yonis H, Argaud L, Heunks L, Louis B. Low-pressure support vs automatic tube compensation during spontaneous breathing trial for weaning. Ann Intensive Care. 2019 Dec 13;9(1):137. doi: 10.1186/s13613-019-0611-y. PMID 31836913
- [Background] El-Shahat, H., Salama, S., Wafy, S. et al. Automatic tube compensation versus pressure support ventilation as a weaning mode: does it make a difference?. Egypt J Bronchol 9, 253-260 (2015). https://doi.org/10.4103/1687-8426.165905
- [Background] Haberthur C, Mols G, Elsasser S, Bingisser R, Stocker R, Guttmann J. Extubation after breathing trials with automatic tube compensation, T-tube, or pressure support ventilation. Acta Anaesthesiol Scand. 2002 Sep;46(8):973-9. doi: 10.1034/j.1399-6576.2002.460808.x. PMID 12190798
- [Background] Cohen J, Shapiro M, Grozovski E, Fox B, Lev S, Singer P. Prediction of extubation outcome: a randomised, controlled trial with automatic tube compensation vs. pressure support ventilation. Crit Care. 2009;13(1):R21. doi: 10.1186/cc7724. Epub 2009 Feb 23. PMID 19236688
- [Background] Cardinal-Fernandez P, Bougnaud J, Cour M, Argaud L, Poole D, Guerin C. Automatic Tube Compensation During Spontaneous Breathing Trials. Respir Care. 2022 Oct;67(10):1335-1342. doi: 10.4187/respcare.09920. Epub 2022 Jun 21. PMID 36137582
- [Background] Guttmann J, Haberthur C, Mols G, Lichtwarck-Aschoff M. Automatic tube compensation (ATC). Minerva Anestesiol. 2002 May;68(5):369-77. PMID 12029248
- [Background] Burns KEA, Wong J, Rizvi L, Lafreniere-Roula M, Thorpe K, Devlin JW, Cook DJ, Seely A, Dodek PM, Tanios M, Piraino T, Gouskos A, Kiedrowski KC, Kay P, Mitchell S, Merner GW, Mayette M, D'Aragon F, Lamontagne F, Rochwerg B, Turgeon A, Sia YT, Charbonney E, Aslanian P, Criner GJ, Hyzy RC, Beitler JR, Kassis EB, Kutsogiannis DJ, Meade MO, Liebler J, Iyer-Kumar S, Tsang J, Cirone R, Shanholtz C, Hill NS; Canadian Critical Care Trials Group. Frequency of Screening and Spontaneous Breathing Trial Techniques: A Randomized Clinical Trial. JAMA. 2024 Dec 3;332(21):1808-1821. doi: 10.1001/jama.2024.20631. PMID 39382222
- [Background] Burns KEA, Sadeghirad B, Ghadimi M, Khan J, Phoophiboon V, Trivedi V, Gomez Builes C, Giammarioli B, Lewis K, Chaudhuri D, Desai K, Friedrich JO. Comparative effectiveness of alternative spontaneous breathing trial techniques: a systematic review and network meta-analysis of randomized trials. Crit Care. 2024 Jun 8;28(1):194. doi: 10.1186/s13054-024-04958-4. PMID 38849936
- [Background] Burns KEA, Khan J, Phoophiboon V, Trivedi V, Gomez-Builes JC, Giammarioli B, Lewis K, Chaudhuri D, Desai K, Friedrich JO. Spontaneous Breathing Trial Techniques for Extubating Adults and Children Who Are Critically Ill: A Systematic Review and Meta-Analysis. JAMA Netw Open. 2024 Feb 5;7(2):e2356794. doi: 10.1001/jamanetworkopen.2023.56794. PMID 38393729
- [Background] Roberts KJ, Goodfellow LT, Battey-Muse CM, Hoerr CA, Carreon ML, Sorg ME, Glogowski J, Girard TD, MacIntyre NR, Hess DR. AARC Clinical Practice Guideline: Spontaneous Breathing Trials for Liberation From Adult Mechanical Ventilation. Respir Care. 2024 Jun 28;69(7):891-901. doi: 10.4187/respcare.11735. PMID 38443142
- [Background] Mart MF, Brummel NE, Ely EW. The ABCDEF Bundle for the Respiratory Therapist. Respir Care. 2019 Dec;64(12):1561-1573. doi: 10.4187/respcare.07235. Epub 2019 Nov 5. PMID 31690615
- [Background] Boles JM, Bion J, Connors A, Herridge M, Marsh B, Melot C, Pearl R, Silverman H, Stanchina M, Vieillard-Baron A, Welte T. Weaning from mechanical ventilation. Eur Respir J. 2007 May;29(5):1033-56. doi: 10.1183/09031936.00010206. PMID 17470624
- [Background] Roberts KJ. 2022 Year in Review: Ventilator Liberation. Respir Care. 2023 Nov 25;68(12):1728-1735. doi: 10.4187/respcare.11114. PMID 37402584
- [Background] Trudzinski FC, Neetz B, Bornitz F, Muller M, Weis A, Kronsteiner D, Herth FJF, Sturm N, Gassmann V, Frerk T, Neurohr C, Ghiani A, Joves B, Schneider A, Szecsenyi J, von Schumann S, Meis J. Risk Factors for Prolonged Mechanical Ventilation and Weaning Failure: A Systematic Review. Respiration. 2022;101(10):959-969. doi: 10.1159/000525604. Epub 2022 Aug 17. PMID 35977525